CLINICAL TRIAL: NCT07028437
Title: The Effect of Endoscopy-assisted Transoral Parotid Gland Tumor Excision Compared With Traditional Operation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Youyuan Wang, Associate Chief Physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSJS-2024-075-02
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Benign Tumor of Parotid Gland; Endoscope-assisted Surgery; Gland Preservation; Minimally Invasive Surgery
Keywords: transoral parotid gland tumor excision; Endoscope-assisted; minimally invasive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic-assisted transoral approach for parotid tumor resection (Experimental): A 5-7 cm curvilinear incision was made with electrocautery on the buccal mucosa along the anterior border of the pterygomandibular raphe on the affected side. The mucosal flap was elevated superiorly, with preservation of the parotid duct and buccal nerve. Two assistants were required to maintain retractor elevation, and hold the endoscope. Electrocautery dissection was performed in three dimensions to expose the anterior borders of both the medial pterygoid muscle and masseter muscle, along with the tumor mass. The surgeon manipulated either electrocautery or ultrasonic scalpel for precise dissection, and used forceps to retract or displace muscular and parotid tissues. Hemoclips were applied to achieve hemostasis. Blunt dissection through normal peri-tumoral tissue ensured complete tumor resection while preserving critical structures including facial nerve branches, buccal nerve, and parotid duct.
  Interventions: Procedure: Endoscopic-assisted transoral approach for parotid tumor resection
- Blair S-shaped incision for parotid tumor (Other): The traditional parotid tumor resection surgery employs a Blair S-shaped incision, starting from the anterior edge of the tragus, extending along the auricle to the earlobe, then curving downward along the posterior border of the mandibular ramus to a point 2-3 cm below the mandibular angle. The skin and subcutaneous tissues are incised to the superficial layer of the parotid fascia, followed by anterior flap elevation while preserving the branches of the greater auricular nerve. The parotid gland and tumor are then exposed, with careful dissection of the facial nerve before removing the tumor and gland. The preservation of critical structures is similar to that in the endoscopic-assisted transoral approach group. A negative-pressure drainage tube is placed at the incision site, and the wound is closed in layers.
  Interventions: Procedure: Blair S-shaped incision for parotid tumor

INTERVENTIONS:
Procedure: Endoscopic-assisted transoral approach for parotid tumor resection — The buccal mucosa was incised in front of the mandibular ligament of the inner wing of the mouth, the submucosal tissue was separated, and important structures such as the buccal nerve, parotid duct, and facial nerve were protected. The tumor was completely resected while preserving the parotid gland.
  Arms: Endoscopic-assisted transoral approach for parotid tumor resection
Procedure: Blair S-shaped incision for parotid tumor — The Blair S-shaped incision was made through an anterior auricular incision. After cutting the skin, the flap was reflapped. The greater auricular nerve and facial nerve were separated and protected, and the tumor was completely resected.
  Arms: Blair S-shaped incision for parotid tumor

SUMMARY:
Endoscopic-assisted surgery has become a popular technique in salivary gland surgery, particularly for parotid gland tumors. However, this technique has not yet been routinely applied to transoral parotid tumor resection. This retrospective study aimed to evaluate the outcomes of gland-preserving surgery in patients with benign parotid tumors undergoing endoscopic-assisted transoral resection.

The study included 30 patients with benign parotid tumors who underwent gland-preserving tumor resection: 15 underwent endoscopic-assisted transoral resection, while the other 15 underwent conventional tumor resection via the Blair S-shaped incision. Surgical feasibility, perioperative variables, postoperative appearance, and functional outcomes were assessed.

In both groups, all tumors were completely removed with negative margins. No significant differences were observed between the two groups in terms of intraoperative blood loss, postoperative drainage volume, average incision length, or facial nerve injury. However, the endoscopic-assisted transoral group demonstrated superior cosmetic outcomes. No tumor recurrence was observed during the 1-6 month follow-up period.

Therefore, endoscopic-assisted transoral parotid tumor resection is a safe approach for benign parotid tumors, offering both favorable functional and aesthetic results.

DETAILED DESCRIPTION:
The incidence of parotid gland tumors is approximately 1 in 100,000, accounting for 80% of all salivary gland tumors, with about 80% being benign. Parotid tumor resection is a well-established surgical technique. Traditionally, the Blair S-shaped incision has been used, but it leaves noticeable scars on the maxillofacial region, which can be a significant burden for both surgeons and patients. Additionally, postoperative complications such as great auricular nerve injury may occur.

In the mid-20th century, the standard surgical approaches for benign parotid tumors included total parotidectomy (with facial nerve sacrifice) or superficial parotidectomy (preserving the facial nerve), which significantly reduced tumor recurrence rates. However, due to the extensive surgical scope, these procedures were associated with a high incidence of complications such as facial nerve dysfunction, Frey's syndrome, salivary fistula, and facial scar deformities.

In recent years, with growing interest in minimally invasive surgery, studies have found that subtotal parotidectomy for benign parotid tumors not only reduces postoperative complications but also maintains comparable recurrence rates. To meet patients' aesthetic demands, more concealed hairline incisions have gained popularity, as the scars can be hidden behind the ear.

With advancements in minimally invasive techniques for parotid tumor surgery, surgeons have developed various approaches to minimize scarring and reduce complications, including retroauricular sulcus incisions, endoscopic-assisted techniques, and transoral/intraoral resections. Endoscopic-assisted techniques leave minimal or hidden scars postoperatively. The combination of intraoral incisions and endoscopy can further conceal surgical scars, reduce patient trauma, and improve satisfaction-without significant complications compared to traditional transcutaneous approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary benign parotid tumors all underwent CT, MRI and ultrasound-guided FNAC examinations of parotid tumors before the operation. All the patients underwent glandular preservation surgery.

Exclusion Criteria:

* The tumor diameter is greater than 6cm, has undergone radiotherapy, is a highly malignant tumor, a tumor invading the skin, and a recurrent tumor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
VAS for aesthetic | 1、3、6 months after surgery
  The assessment of postoperative aesthetics includes the Visual Analogue Scale (VAS); 0-10. 0 indicates a poor result and 10 indicates a good result.
aesthetic | 1、3、6 months after surgery
  The appearance assessment section of the University of Washington Quality of Life Questionnaire (UW-QOL)

SECONDARY OUTCOMES:
Incidence of postoperative complications | 1、3、6 months after surgery
  The proportion of patients with complications such as facial paralysis, salivary fistula, hemorrhage, hematoma, and numbness of the earlobe after the operation among the total number of patients in this group

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China